CLINICAL TRIAL: NCT03608800
Title: Potential Effects of Intermittent Fasting to Gut Microbiota of Metabolic Syndrome Subjects
Brief Title: Potential Effects of Intermittent Fasting to Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Min Xia (Other)
Responsible Party: Sponsor-Investigator, Min Xia, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2018IF01-1
Record Dates: First submitted 2018-07-22; First posted 2018-08-01 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent fasting (Experimental): two nonconsecutive days of 75% diet energy restriction per week for 8 weeks
  Interventions: Behavioral: Intermittent fasting
- Control diet (No Intervention): maintain the energy intake as usual

INTERVENTIONS:
Behavioral: Intermittent fasting — The intervention of two nonconsecutive days of 75% energy restriction per week for 8 weeks
  Arms: Intermittent fasting

SUMMARY:
The survey is designed to investigate whether 8 weeks of discrete two-day intermittent fasting per week will impact gut microbiota and cardiovascular risks of metabolic syndrome subjects.

DETAILED DESCRIPTION:
Intermittent fasting was demonstrated to optimize energy metabolism and promote health. However, the benefits of intermittent fasting to gut microbiota are remain unclear. Further evidence is needed in understanding the effects of intermittent fasting to gut microbiota and cardiovascular risks in subjects with metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* Local residents aged between 30 to 50 years old
* Stable body weight (change <±10% of body weight) for 3 months before the study
* Central obesity: waist circumference ≥90 cm in males or ≥80 cm in females; plus any two of the following four conditions:

  1. Elevated triglycerides: serum triglycerides ≥150 mg/dL (1.7 mmol/L)
  2. Reduced HDL cholesterol: serum HDL-c <40 mg/dL (1.03 mmol/L) in males or <50 mg/dL (1.29 mmol/L) in females
  3. Elevated blood pressure: systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥85 mmHg or receiving medication of hypertension
  4. Elevated fasting plasma glucose: fasting plasma glucose ≥100 mg/dL (5.6 mmol/L)

Exclusion Criteria:

* History of cardiovascular and cerebrovascular diseases
* Acute or chronic infectious diseases within 4 weeks
* Known malignant tumor
* Alcohol abuse (weekly consumption of alcohol is more than 70 g in females or 140 g in males)
* Regular therapy with antihypertensive drug, hypolipidemic agents, hypoglycemic agents, hormonal agents and antidepressants within 6 months
* Use of probiotics, prebiotics or antibiotics within 3 months and in progress of study
* Use of antiinflammatory drug in progress of study
* Following a vegetarian diet or veganism
* Women who are pregnant or intend to be pregnant during the research

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
BMI | 8 weeks
  BMI(weight in kilograms, height in meters and BMI in kg/m^2)
Body fat mass | 8 weeks
  Body fat mass (kg)

SECONDARY OUTCOMES:
systolic pressure | 8 weeks
  systolic pressure(mmHg)
diastolic pressure | 8 weeks
  diastolic pressure(mmHg)
gut microbiota composition | 8 weeks
  gut microbiota composition at different levels of classification determined by 16s rRNA pcr
plasma IL-6 | 8 weeks
  plasma interleukin 6 (pg/mL)
plasma TNF-α | 8 weeks
  plasma TNF-α (pg/mL)
plasma sCD40L | 8 weeks
  plasma soluble CD40 ligand (ng/mL)
plasma leptin | 8 weeks
  plasma leptin (ng/mL)
plasma adiponectin | 8 weeks
  plasma adiponectin (μg/mL)
plasma MDA | 8 weeks
  plasma malondialdehyde (nmol/mL)
plasma oxLDL | 8 weeks
  plasma oxidative LDL (mU/L)
plasma total nitrate | 8 weeks
  plasma total nitrate (mmol/L)
plasma AMDA | 8 weeks
  plasma asymmetric dimethylarginine (ng/mL)
plasma VCAM-1 | 8 weeks
  plasma vascular cell adhesion protein 1 (ng/mL)
plasma vWF | 8 weeks
  plasma Von Willebrand factor (U/mL)
metabolic pathway of gut microbiota | 8 weeks
  metabolic pathway of gut microbiota determined by 16s rRNA pcr

OTHER OUTCOMES:
serum LDL-cholesterol | 8 weeks
  serum LDL-cholesterol(mmol/L);
serum HDL-cholesterol | 8 weeks
  serum HDL-cholesterol (mmol/L);
serum triglyceride | 8 weeks
  serum triglyceride (mmol/L)
serum Apo B/apo A1 | 8 weeks
  serum Apo B/apo A1
serum glucose | 8 weeks
  serum glucose (mmol/L)
serum insulin | 8 weeks
  serum insulin (mU/L)
serum total cholesterol | 8 weeks
  serum total cholesterol (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Min Xia, Doctor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Nutrition and Food Hygiene, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo Y, Luo S, Ye Y, Yin S, Fan J, Xia M. Intermittent Fasting Improves Cardiometabolic Risk Factors and Alters Gut Microbiota in Metabolic Syndrome Patients. J Clin Endocrinol Metab. 2021 Jan 1;106(1):64-79. doi: 10.1210/clinem/dgaa644. PMID 33017844